CLINICAL TRIAL: NCT03810352
Title: Association of Platelet Parameters Identified by the Sysmex XN-1000 and Flow Cytometry With Concurrent and Subsequent Bleeding Severity in Children With Immune Thrombocytopenia (ITP): A Multicenter Study
Brief Title: Association of Platelet Parameters With Bleeding Severity in Children With ITP
Acronym: ITP-APPS
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Sysmex America, Inc. (Industry); Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other); Baylor College of Medicine (Other); Columbia University (Other); Duke University (Other)
Responsible Party: Principal Investigator, Andrew Frelinger, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: P00030227
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; platelet function; Sysmex
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The investigators are using blood samples to measure platelet parameters and biomarkers for platelet function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ITP: Patients with primary or secondary immune thrombocytopenia

SUMMARY:
Patients with severe immune thrombocytopenia (ITP) present with similarly low platelet counts but varying bleeding symptoms, making it difficult to predict the disease course and to decide on an appropriate treatment plan. In a single-center study, platelet parameters including the immature platelet fraction, the absolute immature platelet count , and functional response markers were found to be significantly associated with patient bleeding severity, independent of platelet count. This study aims to confirm and replicate these findings in a multi-center patient population and to investigate the use of these parameters to better predict disease severity and bleeding events.

DETAILED DESCRIPTION:
Many children with severe immune thrombocytopenia (ITP) present with mild symptoms and their disease spontaneously resolves within 3 to 6 months. However, a subset of pediatric ITP patients experience severe bleeds and their symptoms persist for more than 6 to 12 months. Both patient populations present with similarly low platelet counts, making it difficult to predict the disease course and to decide on a treatment plan. The current American Society of Hematology treatment guidelines advise that most cases of ITP may be managed through close observation, while pharmacological interventions that may result in treatment-related toxicities may be used in patients with more severe bleeding symptoms. In order to improve the care and management of pediatric patients with ITP, it is necessary to develop a better predictor of bleeding events and disease severity than the patient's platelet count.

In a previous single-center study, investigators studied the association of different platelet parameters with patient bleeding severity. Using whole blood from patients diagnosed with severe ITP, investigators measured the immature platelet fraction (IPF) and absolute immature platelet count (IPC) through a hematology analyzer (Sysmex XN-1000). Investigators performed functional tests on the platelets and analyzed them through flow cytometry. In this study, the investigators found that the IPF and IPC is associated with patient bleeding severity, independent of platelet count. It was also determined that functional activation markers such as P-selectin and glycoprotein (GP) IIb-IIIa are significantly associated with subsequent bleeding severity in children, independent of platelet count. The results of these proposed studies in ITP patients may suggest clinically relevant uses of these assays.

To confirm these findings, this trial will repeat the previous study in a multi-center patient population, including a greater number of patients with severe bleeding and low platelet counts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary or secondary immune thrombocytopenia.
* Platelet count of < 50 x 10^9/L

Exclusion Criteria:

* May not have received aspirin 10 days prior to study entry.
* May not have received nonsteroidal anti-inflammatory drugs (NSAIDs) 3 days prior to study entry.

Ages: 6 Months to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients diagnosed with primary or secondary immune thrombocytopenia.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-11-26 (Actual)

PRIMARY OUTCOMES:
Association of IPF with concurrent, subsequent and worst-ever bleeding in children with ITP. | February 2019-August 2022
  Evaluate in a multi-center study the association, independent of platelet count, of IPF measured by the Sysmex XN-1000 with concurrent, subsequent, and worst-ever bleeding in children with ITP.
Association of IPC with concurrent, subsequent, and worst-ever bleeding in children with ITP | February 2019-August 2022
  Evaluate in a multi-center study the association, independent of platelet count, of immature platelet parameters measured by the Sysmex XN-1000 (IPC, Plt-F, and FSC and other research parameters as applicable) with concurrent, subsequent, and worst-ever bleeding in children with ITP.
Association of platelet function markers with concurrent, subsequent, and worst-ever bleeding in children with ITP. | February 2019-August 2022
  Evaluate in a multi-center study the association, independent of platelet count, off circulating andd agonist-stimulated platelet surface P-selectin and activated GPIIb-IIIa with concurrent, subsequent, and worst-ever bleeding in children with ITP.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas